CLINICAL TRIAL: NCT00521833
Title: Surgically Induced Astigmatism of Temporal Versus Nasal Clear Corneal Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8380
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-08

CONDITIONS: Surrgical Induced Astigmatism
Keywords: Kataract; Astigmatism; phacoemulsification
MeSH Terms: conditions — Astigmatism | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Temporal (right eye)
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- 2 (Experimental): Nasal (Left eye)
  Interventions: Procedure: phacoemulsification and intraocular lens implantation

INTERVENTIONS:
Procedure: phacoemulsification and intraocular lens implantation — clear cornea phacoemulsification and intraocular lens implantation using temporal or nasal incisions respectively

SUMMARY:
To compare the short-term astigmatic outcomes of phacoemulsification cataract surgery and intraocular lens implantation using temporal versus nasal clear corneal incisions.

DETAILED DESCRIPTION:
In a clinical trial, consecutive eyes with senile cataract underwent phacoemulsification with implantation of a 6.0 mm foldable hydrophobic acrylic intraocular lens through a 3.2 mm horizontal clear cornea incision at 180 degrees (temporal incision in right eyes, nasal incision in left eyes). Keratometric astigmatism was measured preoperatively and one and four weeks and 6 months after surgery. Surgically induced astigmatism (SIA) was calculated by the vector analysis method using the Holladay-Cravy-Koch formula. Patients with history of diabetes mellitus, connective tissue disorders, steroid use, previous ocular surgery, with the rule astigmatism >1D, pseudoexfoliation and any corneal pathology were excluded.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with senile cataract

Exclusion Criteria:

* Previously operated eyes
* Presence of corneal pathology
* Pseudo exfoliation
* With-the-rule (WTR) astigmatism >1 D
* Presence of diabetes mellitus
* History of connective tissue disease
* Consumption of systemic steroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Total and Surgical Induced Astigmatism | At 1 and 4 weeks and 6 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Pakravan, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Ophthalmic research center, Tehran, Tehran Province, Iran